CLINICAL TRIAL: NCT01970605
Title: Silver Graft All Comers Registry is to Assess the Long Term Clinical Benefit of Silver Graft in an Unselected Patient Population
Brief Title: Silver Graft All Comers Registry
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1310
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Aneurysm; Graft Failure; Graft Infection
MeSH Terms: conditions — Aneurysm | interventions — Blood Vessel Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with PAOD or aneurysms: Patients
  * in Fontaine class > IIa,
  * in need of aneurysm repair,
  * with defined cardiovascular risk factors or
  * graft infections.
  Surgical reconstruction with defined Silver Graft vascular prosthesis.
  Interventions: Procedure: Surgical reconstruction

INTERVENTIONS:
Procedure: Surgical reconstruction — In contrast to silver acetate impregnated vascular graft, Silver Graft can be immersed in an antibiotic containing solution prior to implantation. This practice should always be followed according to each participant's hospital guidelines and experience. The long term efficacy of the metallic silver coating will not be reduced.
  Common practice antibiotic co-medication before, during and after surgery needs to be documented but is at the discretion of each participating institution.
  Due to the registry character of this assessment, i.e. routine use of the investigational product, local antibiotics, e.g. dipping of the vascular graft into a rifampin solution is permissible.
  Other Names: Vascular reconstruction; Vascular prosthesis; Silver Graft

SUMMARY:
This web based e-Registry will be international, multi-center and prospective. Silver Graft e-Registry to assess the long term clinical benefit of Silver Graft in an unselected patient population

DETAILED DESCRIPTION:
To assess the long term clinical benefit of Silver Graft in an unselected patient population with Peripheral Artery Occlusive Disease (PAOD) fulfilling one of the the following criteria:

1. Any suitable patient in need of an infrarenal vascular reconstruction with Fontaine class IIb or indicated vascular reconstruction aneurysm repair.

   or
2. Any suitable patient with an increased risk for early graft failure except those mentioned under (3). These may include

   * diabetics
   * Fontaine class> IIb
   * patients of advanced age (≥75 y)
   * patients with renal insufficiency (creatinine ≥ 1.50 mg/dl or ≥130 µmol/l)
   * patients with COPD or documented coronary artery disease (prior PCI, prior CABG, documented myocardial ischemia)
   * patients with major amputation
   * immunosuppressed patients
   * patients with autoimmune disease, malignancy

   or
3. Any suitable patient with graft infection or present infection in the anatomical position of indicated vascular reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Any suitable patient in need of an infrarenal vascular reconstruction with Fontaine class IIb or indicated vascular reconstruction aneurysm repair.
2. Any suitable patient with an increased risk for early graft failure except those mentioned under (3). These may include

   * diabetics
   * Fontaine class> IIb
   * patients of advanced age (≥75 y)
   * patients with renal insufficiency (creatinine ≥ 1.50 mg/dl or ≥130 µmol/l)
   * patients with COPD or documented coronary artery disease (prior PCI, prior CABG, documented myocardial ischemia)
   * patients with major amputation
   * immunosuppressed patients
   * patients with autoimmune disease, malignancy
3. Any suitable patient with graft infection or present infection in the anatomical position of indicated vascular reconstruction.

Exclusion Criteria:

* Any patient with common contraindications for vascular surgery may not be included in this registry.
* Any patient with an estimated life expectancy less than the first follow-up period, i.e. 12 months is excluded from data entry.
* Any patient with a known and documented allergy to silver or silver ions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PAOD Fontaine classification > IIa Patients in need of aneurysm repair Patients in need of revisions, i.e. graft infections
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
graft patency | 12 months
  12-month patency assessed with duplex ultrasound

SECONDARY OUTCOMES:
Freedom from infection | at 12 months
  assessed through clinical parameters, imaging (ultrasound, MRI, CT), bacterial cultures

OTHER OUTCOMES:
Freedom from perigraft fluid presence | 12 months
  assessed through imaging (ultrasound, MRI, CT)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Tautenhahn, MD, Principal Investigator — Klinikum Magdeburg
Locations (1):
- Klinikum Magdeburg, Magdeburg, Germany

REFERENCES:
- [Background] Zegelman M, Guenther G, Waliszewski M, Pukacki F, Stanisic MG, Piquet P, Passon M, Halloul Z, Tautenhahn J, Claey L, Agostinho C, Simici D, Doebrich D, Mueller C, Balzer K. Results from the International Silver Graft Registry for high-risk patients treated with a metallic-silver impregnated vascular graft. Vascular. 2013 Jun;21(3):137-47. doi: 10.1177/1708538113478773. PMID 23508393
- [Background] Zegelman M, Guenther G, Florek HJ, Orend KH, Zuehlke H, Liewald F, Storck M. Results from the first in man german pilot study of the silver graft, a vascular graft impregnated with metallic silver. Vascular. 2009 Jul-Aug;17(4):190-6. doi: 10.2310/6670.2009.00034. PMID 19698298